CLINICAL TRIAL: NCT04683848
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of MT-3921 in Subjects With Acute Traumatic Cervical Spinal Cord Injury
Brief Title: Study to Assess the Efficacy and Safety of MT-3921 in Subjects With Acute Traumatic Cervical Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-3921-A01; jRCT2031210320 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-3921 (Experimental): Intravenous (IV)
  Interventions: Biological: MT-3921
- Placebo (Placebo Comparator): Intravenous (IV)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MT-3921 — Solution for infusion; Intravenous (IV)
  Other Names: Unasnemab
  Arms: MT-3921
Biological: Placebo — Solution for infusion; Intravenous (IV)
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of intravenous (IV) infusions of MT-3921 to placebo in subjects with acute traumatic cervical spinal cord injury.

Subjects meeting eligibility criteria will enter the 6-month double-blind period. Subjects will be randomized in a 2:1 ratio to receive MT-3921 or placebo in a double blind manner.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Provide written informed consent prior to beginning any study procedures
* Cervical spinal cord injury that meet all of the following criteria:

  * Classified as AIS A, AIS B or AIS C
  * ISNCSCI neurological level of injury between C4 and C7 (for C4, the subject must have at least 1 point of motor activity between C5 to C7)
  * UEMS ≤28 at Screening
* Body mass index (BMI) <40

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Any concomitant injury that interferes with the procedures and examinations required by study protocol, including performance, interpretation or validity of neurological examinations
* Poly-traumatic Injury as defined by Injury Severity Score (ISS) values > 25
* Penetrating spinal cord injuries
* Complete transection of the spinal cord
* Any other significant pre-existing medical conditions prior to spinal cord injury or current conditions that, in the judgement of the iInvestigator, may increase the risks associated with study participation
* History of anaphylaxis or clinically significant allergic reactions to any medication
* History or presence of malignancy within the last 3 years prior to screening
* Subjects with current SARS-CoV-2 infection (COVID-19)
* Subjects with hereditary fructose intolerance
* Psychoactive substance use disorder
* Participation in any clinical trial of a new chemical entity within 12 weeks prior to Screening
* Female subjects who are pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Upper Extremity Motor Score (UEMS) | Baseline and at Day 180
  The UEMS is a subscore of the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) that focuses selectively on function of 5 key muscles in the upper limbs. UEMS ranges from 0 to 50 points, where a higher score indicates a better movement.

SECONDARY OUTCOMES:
Change in Spinal Cord Independence Measurement (SCIM) III score | Baseline and at Day 180
  The SCIM III is a comprehensive rating scale that measures the ability of patients with SCI to perform everyday tasks according to their value for the patient. The SCIM III is grouped into four subscales: Self-Care, Respiration and Sphincter Management, Mobility in Room and Toilet, and Mobility Indoors and Outdoors. The total SCIM III score ranges from 0 to 100 points, with 0 point being requiring total assistance and 100 points being completely independent.
Change in Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) score | Baseline and at Day 180
  The GRASSP measures sensorimotor and prehension function through three domains (Strength, Sensation and Prehension) which are important in describing arm and hand function. The total GRASSP score ranges from 0 to 116 points, where a higher score indicates a better outcome.
Change in Spinal Cord Ability Ruler (SCAR) | Baseline and at Day 180
  The SCAR measures voluntary task specific physical actions contributing to independence in ability of daily living. The SCAR uses select items from the upper limb motor assessments of the ISNCSCI and the SCIM III.
Proportion of responders (i.e., subjects with cutoff number or greater increase in the UEMS compared to baseline) | Baseline and at Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (23):
- United States (15):
  - University of California Irvine, Orange, California
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Augusta University, Augusta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Spectrum Health, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis University Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carolinas Rehabilitation, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University - Center for Health & Healing, Portland, Oregon
  - Brooke Army Medical Center in San Antonio, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Carilion Clinic, Roanoke, Virginia
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - NSHA-Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
- Japan (6):
  - Japan Organization of Occupational Health and Safety SPINAL INJURIES CENTER, Izuka-shi, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Hokkaido Spinal Cord Injury Center, Bibai-shi, Hokkaido
  - Japanese Red Cross Kobe Hospital, Kobe, Hyōgo
  - National Hospital Organization Kumamoto Medical Center, Kumamoto, Kumamoto
  - Murayama Medical Center, Musashimurayama-shi, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided